CLINICAL TRIAL: NCT00362388
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy of Intramyocardial Injection of Autologous Bone-Marrow Cells in Patients With Severe, Chronic Ischemic Heart Disease Undergoing Coronary Bypass Surgery
Brief Title: Cell Therapy in Chronic Ischemic Heart Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low enrollling
Sponsor: Ministry of Health, Brazil (Other Government)
Collaborators: Ministry of Science and Technology (Ambiguous)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMRTCC-ISQ
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2008-11

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease
Keywords: Coronary artery disease; Ischemic heart disease; Angiogenesis; Cells; Cardiac surgery
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Intramyocardial injection of autologous bone marrow cells

SUMMARY:
This study was designed to test the hypothesis that direct injection of bone-marrow cells in the heart may increase the number of blood vessels, ameliorating the heart's performance, and relieving patients from symptoms like angina and/or shortness of breath.

DETAILED DESCRIPTION:
Severe ischemic heart disease (IHD) remains a clinical challenge; many patients with IHD have undergone myocardial revascularization procedures (either percutaneous or surgical) but still remain symptomatic despite maximally tolerated medical therapy. Others are considered non-optimal candidates for a complete myocardial revascularization procedure due to the extension and diffuseness of the disease.

Cell therapy with autologous bone marrow-derived cells (BMC) is a novel therapeutic strategy being tested for many cardiovascular diseases, including heart failure, acute myocardial infarction, chronic ischemic heart disease.

The primary objective of this study is to assess the efficacy of intramyocardial injection of autologous BMC on the myocardial perfusion and left ventricular function as an adjunctive therapy (compared to placebo) in patients undergoing coronary artery bypass surgery (CABG).

The secondary objective of this study is to assess the effect of intramyocardial injection of autologous BMC on functional class (angina/heart failure), functional capacity, global and cardiovascular mortality, and quality of life in patients undergoing coronary artery bypass surgery (CABG).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic, severe, diffuse, multivessel atherosclerotic coronary artery disease (CAD) referred for CABG.
* Echocardiogram-assessed LVEF between 25 and 55% (Simpson's rule).
* Angina (or equivalent) functional class II to IV (Canadian Cardiovascular Society) despite maximally tolerated medical therapy.
* Abnormal myocardial perfusion tests:

  i. Cardiac scintigraphy ii. Magnetic resonance imaging iii. Dobutamine-atropine stress-echocardiogram
* Non-candidates for a percutaneous coronary intervention (PCI) due to ANY of the following:

  i. High risk lesion ii. Extensive lesion iii. Diffuse, small vessel disease
* Non-candidates for a complete CABG, or candidates for a complete CABG in whom, according to an expert panel, there is a high probability of failure of the grafts due to the extension and severity of the disease, with diffuse, small vessel involvement.
* To provide a signed, written informed consent, according to the National Guidelines for Clinical Trials.

Exclusion Criteria:

* Severe valve heart disease requiring surgical repair.
* Serologic diagnostic of Chagas' disease.
* Symptoms of heart failure, even from an ischemic etiology, in the absence of objectively documented myocardial ischemia.
* Malignant ventricular arrhythmias (like VT), unless an ICD have been placed.
* Any acute coronary syndrome in the past 3 months.
* End-stage renal disease requiring maintenance dialysis.
* History of neoplasia.
* Drug or alcohol abuse.
* Life expectancy below 2 years.
* Enrollment in any cell therapy trial in the past 2 years.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Reduction in the ischemic score (global/regional) at 12 months; increase in left ventricle ejection fraction (LVEF) at 12 months.

SECONDARY OUTCOMES:
All-cause and cardiovascular mortality during the first year; increase in VO2max, increase in quality of life, reduction in angina/heart failure functional class at 12 months; percentage of patients with a 5% increase in LVEF at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio A. de Oliveira, MD, PhD, Principal Investigator — Heart Institute (InCor), Hospital das Clinicas, University of São Paulo Medical School; Jose Eduardo Krieger, MD, PhD, Study Director — Heart Institute (InCor), Hospital das Clinicas, University of São Paulo Medical School
Locations (6):
- Brazil (6):
  - Irmandade da Santa Casa de Misericórdia, Curitiba, Paraná
  - Clínica Cardiologyca C. Constantini, Curitiba, Paraná
  - Instituto do Coração de Pernambuco do Real Hospital Português de Beneficência, Recife, Pernambuco
  - Instituto Nacional de Cardiologia Laranjeiras (INCL), Rio de Janeiro, Rio de Janeiro
  - Hospital Pró-Cardíaco, Rio de Janeiro, Rio de Janeiro
  - Heart Institute (InCor), Hospital das Clínicas, University of São Paulo Medical School, São Paulo, São Paulo

REFERENCES:
- See also: Link to the Heart Institute (InCor), in São Paulo, Brazil (in Portuguese). — http://www.incor.usp.br
- See also: Link to the Instituto Nacional de Cardiologia Laranjeiras (INCL), in Rio de Janeiro, Brazil (In Portuguese). — http://www.incl.rj.saude.gov.br